CLINICAL TRIAL: NCT00171769
Title: An Open Label, Multi-center Trial to Evaluate the Feasibility and Safety of Short-term Treatment With Subcutaneously Injected Certoparin (8000 U Anti-Xa Twice Daily) in Patients With Persistent Nonvalvular Atrial Fibrillation
Brief Title: Atrial Fibrillation Feasibility Certoparin Trial - AFFECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEX839BDE01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Persistent Nonvalvular Atrial Fibrillation
MeSH Terms: interventions — certoparin

INTERVENTIONS:
Drug: Certoparin

SUMMARY:
This trial is designed to provide data about feasibility and safety of short-term treatment with the low-molecular-weight heparin certoparin in patients with persistent nonvalvular atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* persistent AF (electrical cardioversion is planned)
* written informed consent

Exclusion Criteria:

* acute clinical signs of venous thromboembolism
* current oral anticoagulation
* indication for medical cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-04; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Safety measures including reporting of serious adverse events and adverse events, including vascular and neurological events

CONTACTS AND LOCATIONS:
Overall Officials: novartis pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Result] Tebbe U, Oeckinghaus R, Appel KF, Heuer H, Haake H, Eggers E, Seidel K, Adams J, Harenberg J. AFFECT: a prospective, open-label, multicenter trial to evaluate the feasibility and safety of a short-term treatment with subcutaneous certoparin in patients with persistent non-valvular atrial fibrillation. Clin Res Cardiol. 2008 Jun;97(6):389-96. doi: 10.1007/s00392-008-0644-y. Epub 2008 Mar 5. PMID 18322636